CLINICAL TRIAL: NCT00419939
Title: Improvement of the Interaction Between Motivation, Involvement and Re-learning of Daily Life Competences During the Intensive Neurorehabilitation of Patients With Severe TBI. Development of a Research-based Didactic Model.
Brief Title: Intensive Rehabilitation of Patients With Severe Traumatic Brain Injury - Development of a Didactic Model
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Regionshospitalet Hammel Neurocenter (Other)
Responsible Party: Jørgen Feldbæk Nielsen, Hammel Neurocenter
Other Study IDs: 2007-RHN-01
Record Dates: First submitted 2007-01-08; First posted 2007-01-09 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2011-06

CONDITIONS: Craniocerebral Trauma
Keywords: Severe traumatic brain injury; Intensive neurorehabilitation; "Patient Participation"[Professional-Patient Relations"; Re-learning; Daily life activities; Rehabilitation
MeSH Terms: conditions — Craniocerebral Trauma; Brain Injuries, Traumatic

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: ab 10 patientsr with acquired severe brain injury (GCS 3 - 9), >18 år, PTA phase at the end (GOAT scoring), RLAS score at minimum 4 and informed consent in writing

SUMMARY:
The aim of the study is to develop a research-based pedagogic model to improve the interaction between the patient's motivation, influence and learning.The hypothesis is:

A neuro-rehabilitation effort in patients with severe traumatic brain injury based on a didactic model for improvement of motivation, involvement and re-learning of daily life competences will

* improve the patients experience of meaningful learning and influence
* provide staff with a tool which contributes to the experience to work in a targeted way concerning motivation, patient influence and re-learning daily life competencies

The aim of the study is to develop a research-based didactic model to improve the interaction between the patient's motivation, influence and learning.

DETAILED DESCRIPTION:
Annually, about 7500 people get a traumatic brain injury (TBI) in Denmark. According to Danish and international experiences 250 of these get severe injuries. About 120 younger people often males need highly specialised neuro-rehabilitation at one of the two regional centres in Denmark. Due to the limited amount of research in this field it cannot be documented but assumed, that the patient's motivation and involvement in planning and implementation of rehabilitation improve subjective and objective outcome. Motivation, involvement and learning in patients with severe traumatic brain injury constitute a major challenge. The cases are individual, but often involve disturbances in language and perception, lack of realization, reduced initiative, tiredness and depression. The focus of this project is the intensive physical and psychosocial rehabilitation viewed as a process of relearning targeted daily life competences using the ICF levels of function, activity and participation.

ELIGIBILITY:
Inclusion Criteria:

1. Severe traumatic brain injury (GCS 3-9)
2. Older than 18 years
3. Post Traumatic Amnesiphase (PTA) at the end, 4 Ranchos Los Amigos (RLAS) score at minimum 4
4. Informed consent

Exclusion Criteria:

1. Younger than 18 years
2. In PTA phase
3. RLAS score lower than 4
4. No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ab 10 patientsr with acquired severe brain injury (GCS 3 - 9), >18 år, PTA phase at the end (GOAT scoring), RLAS score at minimum 4 and informed consent in writing
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2007-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Improvement of the patients experience of meaningful learning and influence | 4 -8 weeks

SECONDARY OUTCOMES:
Provide staff with a tool which contributes to the experience to work in a targeted way concerning motivation, patient influence and re-learning daily life competencies | 4 - 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Koch-Jensen, Head of c, Study Director — Regionshospitalet Hammel Neurocenter; Marit Kirkevold, Professor, Study Chair — Department of nursing science, Aarhus University; Lena Aadal, Ph.d stud., Principal Investigator — Regionshospitalet Hammel Neurocenter
Locations (1):
- Regional Hospital Hammel Neurorehabilitation Centre, Voldbyvej 15, Hammel, Denmark